CLINICAL TRIAL: NCT02899858
Title: Restoration of Standing and Walking With ISMS in Humans
Acronym: ISMS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding stopped and no one met IRB approved enrollment criteria
Sponsor: Vanderbilt University (Other)
Collaborators: University of Alberta (Other); Belmont University (Other)
Responsible Party: Principal Investigator, Peter Konrad, MD, PhD, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 140503
Record Dates: First submitted 2016-08-26; First posted 2016-09-14 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injury; Paralysis
Keywords: Thoracic spinal cord injury; Paralysis; ASIA A; Device
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IntraSpinal Micro-Stimulation (Experimental): IntraSpinal Micro-Stimulation will be performed using a maximum of 16 electrodes inserted along each side of spinal cord that correlate with movements created across all 3 joints (hips, knees, and ankles)
  Interventions: Other: Movement Assessment; Other: MRI Scan; Procedure: IntraSpinal Micro-Stimulation; Other: Follow up clinical exam; Other: Post Op MRI Scan; Other: Follow up gait assessment

INTERVENTIONS:
Other: Movement Assessment — Documentation of ASIA A (T2-8) status at Belmont Gait Lab
Other: MRI Scan — Total MRI of spine to evaluate condition of spinal cord
Procedure: IntraSpinal Micro-Stimulation — IntraSpinal Micro-Stimulation will be performed using a maximum of 16 electrodes inserted along each side of spinal cord that correlate with movements created across all 3 joints (hips, knees, and ankles)
Other: Follow up clinical exam — All subjects will be expected to return for a follow-up visit with Drs. Konrad at 1, 3 and 6 month follow up visits.
Other: Post Op MRI Scan — An MRI will be obtained at 3 months following the procedure to document the impact of the mapping procedure on spinal cord anatomy.
Other: Follow up gait assessment — Follow-up assessment with the Belmont Gait Lab will be performed at the 6 month follow up visit

SUMMARY:
Spinal cord neural circuitry exists in the lumbar enlargement that makes it possible to stand and create synergistic, rhythmic stepping activity in the lower limbs. In the past 20 years, clinicians have tried to reengage such these circuits for standing and walking in the lower spinal cord of paralyzed humans through novel paradigms of physical therapy, pharmacological stimulation of the spinal cord, or recently - epidural stimulation of the spinal cord. Although standing and stepping with these maneuvers are rudimentary at best, these human studies offer promise to restore controlled, lower extremity movement to the spinal cord injured (SCI) individual. Evidence from animal data suggests that more focal activation of intraspinal circuitry (IntraSpinal Micro-Stimulation - ISMS) would produce more fatigue resistant, natural standing and stepping activity in humans. To date, there has been no direct confirmation of such circuitry in the spinal cord of bipedal humans who have been paralyzed. Furthermore, mapping of such circuitry would provide the basis of a novel intraspinal neuroprosthetic that should be able to restore control of standing or walking in a manner that is much more physiologically normal and tolerable than by stimulating each individual muscle group. Proof of the existence of these spinal circuits in man, and the ability to activate and control these circuits by first mapping the spinal cord is the basis of this proposal.

DETAILED DESCRIPTION:
Two study volunteers who are completely paralyzed (T2-8 region) to undergo an evaluation of ISMS during an otherwise normal thoracic spinal surgical procedure.

The potential volunteers will be asked to review and sign a screening consent form prior to initial screening. This is to ensure that the ideal two patients are selected for this study and that foreseeable issues are identified and risks minimized for the volunteers. The subjects must have a stable, complete spinal cord injury involving their upper thoracic spinal cord (T2-8 region), and are otherwise planning to undergo a spine surgery involving the lower thoracic spinal cord.

Subjects who have volunteered for this study will undergo their intended spinal surgery by the clinical team. The usual indications for undergoing such a surgery is either to correct a deformity involving the lower thoracic region, or stabilizing the lower thoracic region due to chronic instability from degenerative disease. The surgery intended for clinical treatment must involve exposure of the T9-T12 spinal lamina. However, exposure of the spinal cord through a dural opening would not normally be performed in this clinical scenario. The experimental portion of the surgery begins then, with a laminectomy of T9-T12 and exposure of the spinal cord through a durotomy using standard neurosurgical techniques for spinal cord exposure. The spinal cord in this region will then be mapped and stimulated using ISMS and the effects on the legs measured to determine if the circuitry exists to potentially allow standing or walking through the use of ISMS. The research requests subjects to specifically allow 2 hours of extra time during the routine spinal surgery to perform this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years old; male or female (no preference).
2. Complete paraplegia (ASIA A classification) as a result of a spinal cord injury between the levels of T2-8.

   i. No motor or sensory function below the level of injury as determined by a physician.

   ii. No voluntary bladder function - defined as the inability to sense bladder fullness or voluntary contraction of the bladder (meets criteria for no sacral sparing).

   iii. Stable paraplegia.
3. Patients with involuntary spasms are allowed. However, spasticity must be less than Ashworth 4 or spasm rating of 3 or less.
4. History of spinal cord injury greater than 1 year.
5. Intent to undergo spine surgery involving exposure of at least T9-T12 vertebral lamina.
6. MRI studies performed within the past year showing presence of spinal cord between T8-L1 with reasonable normal anatomical shape. No chronic infections.
7. Ability to travel to Vanderbilt Medical Center.

Exclusion Criteria:

1. Acute medical conditions that are under active treatment. Examples include active urinary tract infection, respiratory illness, decubital ulcers, fractures, upper extremity injury, back pain.
2. Pregnancy.
3. Presence of a neurostimulator, bladder stimulator, cardiac stimulator or other electrical stimulator device implant.
4. Inability to transfer from wheel chair to chair or bed.
5. Inability to tolerate 1 hour of physical activity such as gait training in a harness.
6. Severe depression requiring active medical treatment or counseling.
7. Cognitive impairment that places the study volunteer under the 6th grade reading level.
8. Inability to provide consent.
9. Intradural or extradural masses compressing or displacing the spinal cord between T8-L1 region.
10. Significant change in motor or sensory function over the previous year.
11. History of spinal cord injury less than 1 year.
12. Previous laminectomy and intradural spinal cord procedure involving the region of T9-T12.
13. Patients with involuntary spasms with rigidity more than Ashworth 4 or spasm rating of 3 or more.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
IntraSpinal Micro-Stimulation | 3 years
  Movement of either or both lower extremities while the subject is anesthetized during routine spinal surgery will be performed.

SECONDARY OUTCOMES:
ISMS data collection: | 3 years
  Kinesiology measurement data collected from Dr. Robinson's Gait lab preoperatively will be compared with intraoperative movement data.

OTHER OUTCOMES:
ISMS data review | 3 years
  Human data collected in this study will be compared with pre-clinical animal data from U Alberta, Canada by Dr. Mushahwar's team.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Konrad, MD PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the DSMB when screening and recruiting subjects and when a subject exits the study
Supporting Information: Study Protocol
Time Frame: Within 1 year of closure of study
Access Criteria: Written report of protocol shared with sponsoring agency - US Army.

REFERENCES:
- [Background] Mushahwar VK, Jacobs PL, Normann RA, Triolo RJ, Kleitman N. New functional electrical stimulation approaches to standing and walking. J Neural Eng. 2007 Sep;4(3):S181-97. doi: 10.1088/1741-2560/4/3/S05. Epub 2007 Aug 22. PMID 17873417
- [Background] Bamford JA, Mushahwar VK. Intraspinal microstimulation for the recovery of function following spinal cord injury. Prog Brain Res. 2011;194:227-39. doi: 10.1016/B978-0-444-53815-4.00004-2. PMID 21867807
- Available data/document: Study Protocol: 140503 — https://www4.vanderbilt.edu/irb/